CLINICAL TRIAL: NCT02631538
Title: A Randomized, Double Blind (Sponsor Open), Comparative, Multicenter Study to Evaluate the Safety and Efficacy of Subcutaneous Belimumab (GSK1550188) and Intravenous Rituximab Co-administration in Subjects With Primary Sjögren's Syndrome
Brief Title: Safety and Efficacy Study of Subcutaneous Belimumab and Intravenous Rituximab Co-administration in Subjects With Primary Sjogren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201842; 2015-000400-26 (EudraCT Number)
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Sjogren's Syndrome
Keywords: Subcutaneous; Rituximab; Intravenous; Safety; Efficacy; Sjogren's syndrome; Belimumab
MeSH Terms: conditions — Sjogren's Syndrome | interventions — belimumab; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Subjects will receive belimumab placebo weekly subcutaneous injections to Week 52 and rituximab placebo infusions at Weeks 8 and 10.
  Interventions: Drug: Placebo belimumab; Drug: Placebo rituximab
- Belimumab monotherapy (Experimental): Subjects will receive 200 mg weekly subcutaneous injections of belimumab to Week 52 and placebo rituximab infusions at Weeks 8 and 10.
  Interventions: Drug: Belimumab; Drug: Placebo rituximab
- Belimumab and Rituximab co-administration therapy (Experimental): Subjects will receive belimumab 200 mg SC weekly for 24 weeks followed by weekly placebo belimumab injections to Week 52 with rituximab 1000 mg intravenously at Weeks 8 and 10.
  Interventions: Drug: Belimumab; Drug: Rituximab; Drug: Placebo belimumab
- Rituximab monotherapy (Active Comparator): Subjects will receive 1000 mg IV rituximab infusions at Weeks 8 and 10 and weekly subcutaneous injections of placebo belimumab to Week 52.
  Interventions: Drug: Rituximab; Drug: Placebo belimumab

INTERVENTIONS:
Drug: Belimumab — Belimumab will be provided as a 200 mg sterile, liquid product in a prefilled syringe. Each syringe contains 1.0 mL of 200 mg/mL belimumab. Each syringe will be a single use.
  Arms: Belimumab and Rituximab co-administration therapy; Belimumab monotherapy
Drug: Rituximab — Rituximab will be provided as a 100 mg concentrated solution for infusion. It is a clear, colorless liquid.
  Arms: Belimumab and Rituximab co-administration therapy; Rituximab monotherapy
Drug: Placebo belimumab — The placebo control will be provided as a sterile liquid product in a prefilled syringe. Each syringe will be of a single use.
  Arms: Belimumab and Rituximab co-administration therapy; Placebo; Rituximab monotherapy
Drug: Placebo rituximab — Placebo rituximab will be provided as solution for infusion. It is a clear, colorless liquid.
  Arms: Belimumab monotherapy; Placebo

SUMMARY:
This study is a multi-national, multi-center, double-blind (sponsor open), randomized, placebo-controlled trial in subjects with active primary Sjögren's syndrome designed to understand the safety and tolerability profile of belimumab/ rituximab co-administration and of belimumab monotherapy; and to evaluate whether either co-administration therapy or belimumab monotherapy has a substantive effect on disease activity.

This study will consist screening period, double blind treatment period, a general follow-up period and individualized follow-up period. Approximately 70 subjects will be recruited into the study initially. At Day 0, subjects will be randomized 1:2:2:2 to one of the four treatment arms placebo arm, belimumab monotherapy arm, co-administration therapy arm and rituximab monotherapy arm. Once a sufficient number of subjects have completed the Week 24, interim analyses and sample size re-estimation will be conducted. The total number of subjects randomized may increase following sample size re-estimation up to a maximum of 120 recruited into the study.

Subjects in all arms will receive investigational product (IP) until Week 52 (completion of the treatment phase). All subjects will enter a 16-week general follow-up period after the Week 52 visit or after discontinuation if a subject discontinues IP and withdraws from the treatment phase visits prior to Week 52.

After completing the general follow-up period, subjects with cluster of differentiation (CD)19+ B-cell levels below the lower limit of normal (or less than 90 percent [%] of baseline, if baseline value was below lower limit of normal [LLN]) will enter an individualized safety follow-up phase and return to the clinic for visits every 12 weeks with monthly calls between visits to evaluate subjects for any serious adverse events (SAEs) related to IP or study participation, fatal SAEs, and designated adverse event of special interests (AESIs) (i.e., infections, malignancies, or depression, suicide/self-injury), and to check concomitant medications.

The total duration of participation of a subject in this study will be approximately up to a maximum of 2 years (i.e., up to Week 104).

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years, at the time of signing the informed consent.
* Documented Primary Sjögren's Syndrome by American European Consensus Group criteria including: either anti-Sjogren's-syndrome-related antigen A (SS-A) or anti-Sjogren's-syndrome-related antigen B (SS-B) positive.
* Baseline unstimulated salivary flow >0.0 mL/min or evidence of glandular reserve function (stimulated baseline salivary flow >0.05 mL/min).
* Symptomatic oral dryness (>=5/10 on subject completed numeric response scale).
* Systemically active disease, ESSDAI >=5 points.
* Male and female subjects; females of child bearing potential are eligible if using effective contraception: Female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotropin [hCG] test), not lactating, and at least one of the following conditions applies:

  1. Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy.

     Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study; otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
  2. Reproductive potential and agrees to follow one of the options in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication up to Week 68 after Day 0.
* Ability to understand and comply with the protocol-required procedures and provision of informed consent.

Exclusion Criteria:

* Diagnosis of secondary Sjögren's syndrome.
* Active life-threatening or organ-threatening complications of Sjogren's-syndrome (SS) disease at the time of screening based on treating physician evaluation including but not restricted to (1) vasculitis with renal, digestive, cardiac, pulmonary or central nervous system (CNS) involvement characterized as severe, (2) active CNS or peripheral nervous system (PNS) involvement requiring high dose steroids, (3) severe renal involvement defined by objective measures, (4) lymphoma.
* History of major organ transplant (including hematopoietic stem cell transplant).
* History of malignancy within past 5 years (with the exception of adequately treated: [1] cervical carcinoma Stage 1B or less, [2] non-invasive basal cell and squamous cell skin carcinoma).
* History of infection requiring long term systemic therapy including: (1) history of positive human immunodeficiency virus (HIV) serology, (2) positive serology for Hepatitis C virus (HCV), (3) positive serology for Hepatitis B (HB), defined as: HB surface antigen positive (HBsAg+) OR HB core antibody positive (HBcAb+).
* Previous serious opportunistic or atypical infections or hospitalization for treatment of infection within 364 days of Day 0 or use of parenteral (intravenous [IV] or intramuscular [IM]) antibacterials, antivirals, anti-fungals, or anti-parasitic agents within 364 days of prior to Day 0.
* Patients in a severely immunocompromised state.
* History of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
* History of significant medical illness (or planned surgical procedure) which in the opinion of the investigator would interfere with the study procedures and / or assessments - including but not limited to immunoglobulin G4 (IgG4) disease or prior head or neck irradiation.
* Severe heart failure (New York Heart Association, Class IV) or other severe, uncontrolled cardiac disease.
* Tuberculosis (TB), defined as: prior history of TB infection; suspicion of TB infection or current TB infection
* At risk of suicide, as indicated by a lifetime history of attempted suicide or significant suicidal ideation over the 6 months prior to the screening visit; or, if in the Investigator's judgment, the subject is at risk for a suicide attempt.
* Neurological findings consistent with Progressive Multifocal Leukoencephalopathy (PML) - not otherwise explained - or confirmed PML.
* Electrocardiogram (ECG) showing a clinically significant abnormality at Screening or showing an average corrected QT using Bazett's formula (QTcB) or corrected QT using Fridericia's formula (QTcF) interval >=450 milliseconds (msec) (>=480 msec for subjects with a Bundle Branch Block) over 3 consecutive ECGs.
* Alanine aminotransferase (ALT) >2x upper limit of normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Use of systemic immunosuppressive or immunomodulatory agents including methotrexate, azathioprine, leflunomide, mycophenolate (including mycophenolate mofetil, mycophenolate mofetil hydrochloride, and mycophenolate sodium), mizoribine, calcineurin inhibitors [e.g., tacrolimus, cyclosporine], sirolimus, 6-mercaptopurine, or thalidomide within 60 days prior to Day 0.
* Have received cyclophosphamide within 180 days prior to Day 0.
* Have received anti- B lymphocyte stimulator (BLyS), anti-CD 20, anti-CD22 or anti-CD52 or any other B-cell depleting agent within 364 days prior to Day 0.
* Have received abatacept or any biologic agent within 180 day prior to Day 0 (with exception of denosumab).
* Have received intravenous immunoglobulin (IVIG) or plasmapheresis within 90 days prior to Day 0.
* Have received oral steroid >10 milligram (mg) prednisone equivalent/day within 30 days prior to Day 0 or oral steroid >20 mg prednisone equivalent / day for a minimum of two consecutive weeks within 60 days prior to Day 0. Have received parenteral steroid within 60 days prior to Day 0.
* Have received a live vaccine within 30 days of Day 0.
* Current participation in any other interventional trial.
* Planned blood donation during the treatment and follow up periods of the study.
* Subjects who are unable or unwilling to administer, or to have a caregiver administer subcutaneous injections.
* Drug or alcohol abuse or dependence.
* History of hypersensitivity to belimumab and/or rituximab or known to have titers of human anti-mouse antibody or human anti-chimeric antibody or history of hypersensitivity reactions when treated with other diagnostic or therapeutic monoclonal antibodies.
* Have an IgA deficiency (IgA level <10 milligram per deciliter [mg/dL]).
* Any of the following screening laboratory values: White blood cells (WBC) <2 x 10^9/L; Neutrophils <1.5 x 10^9/Liter (L); Circulating IgG or IgM levels <lower limit of normal (according to central laboratory range); Aspartate aminotransferase (AST) >2.0 times the upper limit of normal; Alkaline phosphatase (ALP) >1.5 times the upper limit of normal; Bilirubin >1.5 times the upper limit of normal; CD4 count <400 cells per cubic millimetre (cells/mm^3); CD8 count <150 cells/mm^3; CD19+ B-lymphocyte counts <0.1 x 10^9/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- Argentina (2):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Trois-Rivières, Quebec
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
- Germany (5):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Bad Abbach
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (5):
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Padua
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Rotterdam
- GSK Investigational Site, Oslo, Norway
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
- Sweden (2):
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Stockholm
- United Kingdom (4):
  - GSK Investigational Site, Swindon, Wiltshire
  - GSK Investigational Site, Edgbaston
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mariette X, Barone F, Baldini C, Bootsma H, Clark KL, De Vita S, Gardner DH, Henderson RB, Herdman M, Lerang K, Mistry P, Punwaney R, Seror R, Stone J, van Daele P, van Maurik A, Wisniacki N, Roth DA, Tak PP. A randomized, phase II study of sequential belimumab and rituximab in primary Sjogren's syndrome. JCI Insight. 2022 Dec 8;7(23):e163030. doi: 10.1172/jci.insight.163030. PMID 36477362
- [Derived] Raymond K, Maher S, Saucier CD, O'Connor M, Yarlas A, Kosinski M, Chen WH, Gairy K. Validation of the PROFAD-SSI-SF in Patients with Primary Sjogren's Syndrome with Organ Involvement: Results of Qualitative Interviews and Psychometric Analyses. Rheumatol Ther. 2023 Feb;10(1):95-115. doi: 10.1007/s40744-022-00493-2. Epub 2022 Oct 13. PMID 36227531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 10 countries across 31 centers. Participants were randomized to receive one of the four treatments; Placebo, Belimumab + Rituximab Co-administration therapy, Belimumab Monotherapy or Rituximab Monotherapy.
Pre-assignment Details: A total of 162 participants were screened of which 76 were screen failures. A total of 86 participants were enrolled in this study.
Groups:
- Placebo: Participants received belimumab matching placebo weekly subcutaneous injections up to Week 52 and rituximab matching placebo infusions at Weeks 8 and 10 in the treatment period. Participants then entered in a 16-week no-treatment General Follow-Up (GFU) period.
- Belimumab + Rituximab Co-administration Therapy: Participants received belimumab 200 milligrams (mg) weekly subcutaneous injections for 24 weeks followed by belimumab matching placebo injections weekly up to Week 52; along with rituximab 1000 mg intravenous infusions at Weeks 8 and 10 in the treatment period. Participants then entered in a 16-week no-treatment GFU period.
- Belimumab Monotherapy: Participants received 200 mg weekly subcutaneous injections of belimumab up to Week 52 and rituximab matching placebo infusions at Weeks 8 and 10 in the treatment period. Participants then entered in a 16-week no-treatment GFU period.
- Rituximab Monotherapy: Participants received 1000 mg intravenous rituximab infusions at Weeks 8 and 10 and weekly subcutaneous injections of belimumab matching placebo up to Week 52 in the treatment period. Participants then entered in a 16-week no-treatment GFU period.
Period: Treatment Period (Up to Week 52)
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy
Started | 13 | 24 | 24 | 25
Completed | 9 | 17 | 19 | 17
Not Completed | 4 | 7 | 5 | 8
Not completed — Adverse Event | 1 | 5 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 5
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Reached stopping criteria | 0 | 0 | 1 | 0
Period: General Follow-up (GFU) (Up to Week 68)
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy
Started | 9 | 17 | 19 | 17
Completed | 8 | 17 | 19 | 16
Not Completed | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy | Total
Number analyzed (Participants) | 13 | 24 | 24 | 25 | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.7 (12.67) | 45.1 (10.93) | 52.0 (11.49) | 55.2 (15.07) | 51.1 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 22 | 22 | 23 | 80
  Male | 0 | 2 | 2 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 2 | 2 | 1 | 6
  American Indian or Alaskan Native | 0 | 0 | 0 | 1 | 1
  Asian - East Asian Heritage | 0 | 1 | 1 | 2 | 4
  White - Arabic/North African Heritage | 0 | 2 | 3 | 0 | 5
  White-White/Caucasian/European Heritage | 12 | 18 | 18 | 21 | 69
  African American/African Heritage and Asian Heritage | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAE) and Non-serious AEs (Non-SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations based on medical or scientific judgment and is associated with liver injury and impaired liver function. Data for number of participants with SAE and non-SAE has been summarized.
Time Frame: Up to Week 68
Population: Safety Population comprised of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy
Number analyzed (Participants) | 13 | 24 | 24 | 25
Participants
  Any SAE | 0 | 3 | 2 | 4
  Any non-SAE | 12 | 24 | 23 | 17

2. Primary Outcome: Number of Participants With Adverse Event of Special Interests (AESIs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AESIs were Malignant Neoplasms, Post-Administration Systemic Reactions (PASR), All Infections of Special Interest (opportunistic infections, herpes zoster, tuberculosis and sepsis), Depression/suicide/self-injury, Deaths and study specific AESI which includes: severe skin reaction per GlaxoSmithKline (GSK) Adjudication, cardiac disorders, Posterior Reversible Encephalopathy Syndrome (PRES) and Progressive multifocal leukoencephalopathy (PML). Data for number of participants with AESI has been summarized.
Time Frame: Up to Week 68
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy
Number analyzed (Participants) | 13 | 24 | 24 | 25
Participants
  Malignant Neoplasms | 0 | 0 | 0 | 1
  PASR | 4 | 2 | 3 | 5
  All Infections of Special Interest | 2 | 1 | 3 | 2
  Depression/Suicide/Self-injury | 0 | 3 | 5 | 1
  Deaths | 0 | 1 | 0 | 0
  Severe Skin Reactions | 0 | 0 | 0 | 0
  Cardiac Disorders | 0 | 1 | 0 | 1
  PRES | 0 | 0 | 0 | 0
  PML | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in European League Against Rheumatism (EULAR) Sjogren's Syndrome Disease Activity Index (ESSDAI) Total Scores Over Time
Description: The ESSDAI is a physician assessed disease activity index developed by EULAR consortium consisting of twelve different clinically relevant organ specific domains; cutaneous, respiratory, renal, articular, muscular, peripheral nervous system, central nervous system, hematological, glandular, constitutional, lymphadenopathy and biological. Each domain has 3 or 4 possible activity levels (i.e., no, low, moderate, high [if available]) using a 4-point scale, ranging from 0 (No activity) to 3 (High activity). Higher score indicates high disease activity. Each domain is assigned a weight between 1 and 6. The Total ESSDAI Scores are obtained by multiplying the level of activity (domain score) by the domain weights, ranges between 0 (no activity) and 123 (highest activity). Higher score indicates more disease activity. Baseline value is the screening visit value (within 35 days prior to Day 0). Change from Baseline was defined as the post-dose visit value minus Baseline value.
Time Frame: Baseline (Screening [within 35 days prior to Day 0]), Week 12, Week 24, Week 36, Week 52 and Week 68
Population: Completer Population comprised of participants who completed the 52 Week treatment visits and general follow up phase of the study including the visit at Week 68. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy
Number analyzed (Participants) | 8 | 17 | 19 | 16
Scores on a scale
  Week 12; n=8, 17, 19 ,15: number analyzed (Participants) | 8 | 17 | 19 | 15
  Week 12; n=8, 17, 19 ,15 | -2.00 (1.449) | -4.85 (0.996) | -3.87 (0.949) | -4.22 (1.048)
  Week 24; n=8, 17, 19 ,16 | -2.87 (1.324) | -5.32 (0.911) | -3.87 (0.869) | -5.25 (0.940)
  Week 36; n=8, 17, 19 ,16 | -3.12 (1.520) | -4.09 (1.045) | -4.23 (0.995) | -4.94 (1.079)
  Week 52;n=8, 17, 19 ,16 | -2.87 (1.294) | -5.67 (0.890) | -4.76 (0.850) | -4.32 (0.919)
  Week 68;n=8, 17, 19 ,16 | -1.75 (1.400) | -5.73 (0.962) | -3.87 (0.918) | -4.38 (0.994)
Statistical Analysis 1: Comparison: Placebo vs Belimumab + Rituximab Co-administration Therapy; Test type: Other; Least square (LS) mean difference = -2.86, 95% CI 2-sided [-6.38 to 0.67], Standard Error of Mean 1.758 — Week 12. Analysis was performed using mixed effects repeated measures model, with Baseline, treatment, visit and interactions of visit with treatment as fixed effects and participant as a random effect
Statistical Analysis 2: Comparison: Belimumab + Rituximab Co-administration Therapy vs Belimumab Monotherapy; Test type: Other; LS mean difference = -0.99, 95% CI 2-sided [-3.75 to 1.78], Standard Error of Mean 1.382 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Belimumab + Rituximab Co-administration Therapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = -0.63, 95% CI 2-sided [-3.52 to 2.26], Standard Error of Mean 1.442 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Belimumab Monotherapy; Test type: Other; LS mean difference = -1.87, 95% CI 2-sided [-5.34 to 1.60], Standard Error of Mean 1.732 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Belimumab Monotherapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = 0.35, 95% CI 2-sided [-2.50 to 3.20], Standard Error of Mean 1.422 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Belimumab + Rituximab Co-administration Therapy; Test type: Other; LS mean difference = -2.45, 95% CI 2-sided [-5.67 to 0.77], Standard Error of Mean 1.607 — Week 24. Analysis was performed using mixed effects repeated measures model, with Baseline, treatment, visit and interactions of visit with treatment as fixed effects and participant as a random effect
Statistical Analysis 7: Comparison: Belimumab + Rituximab Co-administration Therapy vs Belimumab Monotherapy; Test type: Other; LS mean difference = -1.46, 95% CI 2-sided [-3.99 to 1.08], Standard Error of Mean 1.265 — [estimate comment as in outcome 3, analysis 6]
Statistical Analysis 8: Comparison: Belimumab + Rituximab Co-administration Therapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = -0.07, 95% CI 2-sided [-2.68 to 2.55], Standard Error of Mean 1.305 — [estimate comment as in outcome 3, analysis 6]
Statistical Analysis 9: Comparison: Placebo vs Belimumab Monotherapy; Test type: Other; LS mean difference = -1.00, 95% CI 2-sided [-4.17 to 2.18], Standard Error of Mean 1.584 — [estimate comment as in outcome 3, analysis 6]
Statistical Analysis 10: Comparison: Belimumab Monotherapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = 1.39, 95% CI 2-sided [-1.20 to 3.97], Standard Error of Mean 1.290 — [estimate comment as in outcome 3, analysis 6]
Statistical Analysis 11: Comparison: Placebo vs Belimumab + Rituximab Co-administration Therapy; Test type: Other; LS mean difference = -0.97, 95% CI 2-sided [-4.66 to 2.73], Standard Error of Mean 1.845 — Week 36. Analysis was performed using mixed effects repeated measures model, with Baseline, treatment, visit and interactions of visit with treatment as fixed effects and participant as a random effect
Statistical Analysis 12: Comparison: Belimumab + Rituximab Co-administration Therapy vs Belimumab Monotherapy; Test type: Other; LS mean difference = 0.15, 95% CI 2-sided [-2.76 to 3.05], Standard Error of Mean 1.449 — [estimate comment as in outcome 3, analysis 11]
Statistical Analysis 13: Comparison: Belimumab + Rituximab Co-administration Therapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = 0.85, 95% CI 2-sided [-2.15 to 3.86], Standard Error of Mean 1.498 — [estimate comment as in outcome 3, analysis 11]
Statistical Analysis 14: Comparison: Placebo vs Belimumab Monotherapy; Test type: Other; LS mean difference = -1.11, 95% CI 2-sided [-4.76 to 2.53], Standard Error of Mean 1.817 — [estimate comment as in outcome 3, analysis 11]
Statistical Analysis 15: Comparison: Belimumab Monotherapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = 0.71, 95% CI 2-sided [-2.25 to 3.66], Standard Error of Mean 1.476 — [estimate comment as in outcome 3, analysis 11]
Statistical Analysis 16: Comparison: Placebo vs Belimumab + Rituximab Co-administration Therapy; Test type: Other; LS mean difference = -2.80, 95% CI 2-sided [-5.95 to 0.34], Standard Error of Mean 1.570 — Week 52. Analysis was performed using mixed effects repeated measures model, with Baseline, treatment, visit and interactions of visit with treatment as fixed effects and participant as a random effect
Statistical Analysis 17: Comparison: Belimumab + Rituximab Co-administration Therapy vs Belimumab Monotherapy; Test type: Other; LS mean difference = -0.91, 95% CI 2-sided [-3.39 to 1.56], Standard Error of Mean 1.237 — [estimate comment as in outcome 3, analysis 16]
Statistical Analysis 18: Comparison: Belimumab + Rituximab Co-administration Therapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = -1.36, 95% CI 2-sided [-3.91 to 1.20], Standard Error of Mean 1.275 — [estimate comment as in outcome 3, analysis 16]
Statistical Analysis 19: Comparison: Placebo vs Belimumab Monotherapy; Test type: Other; LS mean difference = -1.89, 95% CI 2-sided [-4.99 to 1.21], Standard Error of Mean 1.548 — [estimate comment as in outcome 3, analysis 16]
Statistical Analysis 20: Comparison: Belimumab Monotherapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = -0.44, 95% CI 2-sided [-2.97 to 2.08], Standard Error of Mean 1.261 — [estimate comment as in outcome 3, analysis 16]
Statistical Analysis 21: Comparison: Placebo vs Belimumab + Rituximab Co-administration Therapy; Test type: Other; LS mean difference = -3.99, 95% CI 2-sided [-7.39 to -0.58], Standard Error of Mean 1.699 — Week 68. Analysis was performed using mixed effects repeated measures model, with Baseline, treatment, visit and interactions of visit with treatment as fixed effects and participant as a random effect
Statistical Analysis 22: Comparison: Belimumab + Rituximab Co-administration Therapy vs Belimumab Monotherapy; Test type: Other; LS mean difference = -1.87, 95% CI 2-sided [-4.54 to 0.81], Standard Error of Mean 1.336 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 23: Comparison: Belimumab + Rituximab Co-administration Therapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = -1.35, 95% CI 2-sided [-4.12 to 1.41], Standard Error of Mean 1.379 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 24: Comparison: Placebo vs Belimumab Monotherapy; Test type: Other; LS mean difference = -2.12, 95% CI 2-sided [-5.47 to 1.23], Standard Error of Mean 1.674 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 25: Comparison: Belimumab Monotherapy vs Rituximab Monotherapy; Test type: Other; LS mean difference = 0.51, 95% CI 2-sided [-2.21 to 3.24], Standard Error of Mean 1.362 — [estimate comment as in outcome 3, analysis 21]

4. Secondary Outcome: Stimulated Salivary Flow Rate Over Time
Description: Participants were instructed to chew a piece of paraffin wax for a period of 5 minutes and saliva was collected. The volume of saliva (milliliter) was divided by the duration of the test (minutes) to calculate the stimulated salivary flow rate (milliliter per minute). Baseline value is the screening visit value (within 35 days prior to Day 0).
Time Frame: Baseline (Screening [within 35 days prior to Day 0]), Week 12, Week 24, Week 36, Week 52 and Week 68
Population: Completer Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Milliliter per minute
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy
Number analyzed (Participants) | 8 | 17 | 19 | 16
Milliliter per minute
  Baseline (Screening); n=8, 17, 19 ,16 | 0.470 (0.2470) | 0.714 (0.6294) | 0.425 (0.3292) | 0.618 (0.6211)
  Week 12; n=8, 17, 19 ,16 | 0.486 (0.2045) | 0.754 (0.8342) | 0.493 (0.3733) | 0.581 (0.5265)
  Week 24; n=8, 17, 19 ,16 | 0.554 (0.3054) | 0.784 (0.7900) | 0.454 (0.4105) | 0.724 (0.8901)
  Week 36; n=8, 17, 19 ,15: number analyzed (Participants) | 8 | 17 | 19 | 15
  Week 36; n=8, 17, 19 ,15 | 0.404 (0.2497) | 1.039 (1.1027) | 0.506 (0.4261) | 0.689 (0.5907)
  Week 52; n=8, 17, 19 ,16 | 0.531 (0.3782) | 0.999 (1.1457) | 0.582 (0.6084) | 0.693 (0.7813)
  Week 68; n=8, 17, 19 ,15: number analyzed (Participants) | 8 | 17 | 19 | 15
  Week 68; n=8, 17, 19 ,15 | 0.361 (0.1628) | 0.879 (0.8167) | 0.517 (0.4499) | 0.733 (0.7850)

5. Secondary Outcome: Oral Dryness Numeric Response Scale (NRS) Over Time
Description: Oral dryness was reported by participants on a numeric response scale, ranging from 0 (no dryness) to 10 (maximal dryness), higher score indicates worst imaginable dryness. Baseline value is the screening visit value (within 35 days prior to Day 0).
Time Frame: Baseline (Screening [within 35 days prior to Day 0]), Week 12, Week 24, Week 36, Week 52 and Week 68
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy
Number analyzed (Participants) | 8 | 17 | 19 | 16
Scores on a scale
  Baseline (Screening); n= 8, 17, 19, 16 | 7.6 (1.51) | 7.4 (1.46) | 7.2 (2.14) | 7.3 (1.91)
  Week 12; n=8, 17, 19, 16 | 6.1 (2.59) | 5.7 (1.96) | 6.9 (2.32) | 5.1 (2.77)
  Week 24; n=8, 17, 19, 15: number analyzed (Participants) | 8 | 17 | 19 | 15
  Week 24; n=8, 17, 19, 15 | 5.8 (2.38) | 5.3 (1.83) | 6.8 (2.51) | 5.6 (2.72)
  Week 36; n=8, 17, 19, 16 | 5.8 (2.76) | 5.9 (2.26) | 6.6 (2.19) | 6.2 (2.51)
  Week 52; n=8, 17, 19, 16 | 5.6 (2.13) | 5.7 (1.92) | 7.0 (2.40) | 6.3 (2.32)
  Week 68; n=8, 17, 19, 16 | 6.6 (2.26) | 6.1 (2.63) | 6.9 (2.34) | 6.1 (2.62)

6. Secondary Outcome: Absolute Values for B-cells (Cluster of Differentiation 20 [CD20]) Within Salivary Gland Biopsy at Week 24
Description: Minor salivary gland biopsies were taken for histological analysis to quantify CD20 B Cells.
Time Frame: At Week 24
Population: Completer Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per millimeter square
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy
Number analyzed (Participants) | 8 | 10 | 15 | 12
Cells per millimeter square | 380.21719 (569.908102) | 8.65550 (20.199794) | 396.86058 (781.245844) | 650.76069 (1311.360352)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected up to Week 68.
Description: Safety Population was used to assess SAEs and non-SAEs which comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo | Belimumab + Rituximab Co-administration Therapy | Belimumab Monotherapy | Rituximab Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/24 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/13 | 3/24 | 2/24 | 4/25
Other Adverse Events (participants affected / at risk) | 12/13 | 24/24 | 23/24 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Belimumab + Rituximab Co-administration Therapy (N=24) | Belimumab Monotherapy (N=24) | Rituximab Monotherapy (N=25)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Belimumab + Rituximab Co-administration Therapy (N=24) | Belimumab Monotherapy (N=24) | Rituximab Monotherapy (N=25)
Nasopharyngitis (Infections and infestations) | 4 (10) | 8 (11) | 6 (9) | 3 (4)
Urinary tract infection (Infections and infestations) | 3 (4) | 5 (7) | 3 (9) | 2 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (3) | 3 (4) | 2 (3) | 5 (6)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 3 (4) | 0 (0) | 4 (4) | 1 (2)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 3 (4)
Pneumonia (Infections and infestations) | 2 (2) | 2 (3) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (5) | 6 (6) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Asthenia (General disorders) | 2 (4) | 2 (2) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (10) | 7 (12) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2) | 5 (5) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 5 (7) | 4 (5) | 6 (7)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 6 (9) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (5) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 3 (3) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3) | 1 (1) | 1 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT02631538/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT02631538/SAP_001.pdf